CLINICAL TRIAL: NCT05853549
Title: A Prospective Study to Evaluated the Clinical Implementation Value of an Optical Surface Monitoring System in the Radiotherapy Setup for Patients With Vulvar Cancer, Compared to Standard Laser-based Setup
Brief Title: Clinical Implementation of Surface-guided Radiation Therapy in Vulvar Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pumch-OSMS
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-03

CONDITIONS: Vulvar Cancer
Keywords: Vulvar cancer; Setup error; Intensity-modulated radiation therapy; Optical surface monitoring system
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- optical surface monitoring system group (Experimental): Every radiotherapy fraction from each patients with OSMS technology. Marks were placed on each patient's skin to align the room lasers for presetup, and the setup was completed with information from the OSMS. The deviation values of setup were obtained. The absolute values of setup error and error distribution of the standard laser-based setup and OSMS in the multi-directions were compared.
  Interventions: Device: optical surface monitoring system

INTERVENTIONS:
Device: optical surface monitoring system — An optical surface monitoring system (OSMS) could achieve continuous monitoring of patient position through a nonradiographic and noninvasive technology, which has been widely applied to many sites of radiation therapy, including breast, intracranial, head and neck, abdomen, and extremities

SUMMARY:
This prospective study evaluated the clinical implementation value of an optical surface monitoring system (OSMS) in the radiotherapy setup for patients with vulvar cancer, compared to standard laser-based setup

DETAILED DESCRIPTION:
This was a prospective single-centre trial to investigate the value of OSMS, and we hypothesized that using OSMS would reduce setup error in vulvar cancer treatment compared to a standard laser-based setup. A dose of 45 Gy was delivered to the clinical target volume with intensity-modulated radiation therapy (IMRT) for a total of 25 fractions, followed by 16 to 24 Gy of local electron beam supplementation. Marks were placed on each patient's skin to align the room lasers for presetup, and the setup was completed with information from the OSMS. The deviation values in three translation directions, lateral (Lat), longitudinal (Lng), and vertical (Vrt), and three rotation directions, Rtn (rotation along the z-axis), Pitch (rotation along the x-axis), and Roll (rotation along the y-axis) were obtained. The absolute values of setup error and error distribution of the standard laser-based setup and OSMS were compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be informed of the investigational nature of this study and give written informed consent before treatment.
2. Age ≥18 years and ≤ 85 years.
3. Patients with histologically confirmed vulvar cancer.
4. No evidence of distant metastasis on CT, MRI or positron emission tomograph (PET)/CT.
5. No contraindications to CT scanning.
6. Indications for radiotherapy for vulvar cancer.
7. Adequate marrow: neutrophile granulocyte count ≥1.5*10^9/L, hemoglobin ≥ 80 g/L, platelet count ≥100*10^9/L.
8. Normal liver and kidney function: Creatinine (Cr) < 1.5 mg/dl, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 2*upper limit of normal (ULN).

Exclusion Criteria:

1. No pathological diagnosis.
2. Remote metastasis.
3. Anticipated intolerance of pelvic radiotherapy.
4. Any severe disease which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control, and emotional disturbance.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
The absolute values of setup error | Through study completion, total an average of eight month
  Marks were placed on each patient's skin to align the room lasers for presetup, and the setup was completed with information from the OSMS. The deviation values in multi-directions were obtained. The absolute values of setup error of the standard laser-based setup and OSMS in the above six directions were compared.
The distribution of setup error | Through study completion, total an average of eight month
  Marks were placed on each patient's skin to align the room lasers for presetup, and the setup was completed with information from the OSMS. The deviation values in multi-directions were obtained. The distribution of the standard laser-based setup and OSMS in the above six directions were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Fuquan Zhang, M.D., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Hoisak JDP, Pawlicki T. The Role of Optical Surface Imaging Systems in Radiation Therapy. Semin Radiat Oncol. 2018 Jun;28(3):185-193. doi: 10.1016/j.semradonc.2018.02.003. PMID 29933878